CLINICAL TRIAL: NCT02889861
Title: An Open-label, Multi-center, Rollover Study in Patients With Advanced Melanoma After Completing an IMCgp100 Clinical Study
Brief Title: IMCgp100-401 Rollover Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMCgp100-401
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Malignant Melanoma
Keywords: Uveal melanoma; Cutaneous melanoma
MeSH Terms: conditions — Melanoma; Uveal Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Regimen 1 (Experimental): IMCgp100 (77 kDa bi-specific protein) weekly dosing regimen (QW)
  Interventions: Drug: IMCgp100

INTERVENTIONS:
Drug: IMCgp100 — Bispecific soluble human leukocyte antigen-A2 (HLA-A2) restricted gp100-specific TCR fused to anti-CD3

SUMMARY:
IMCgp100-401 is a rollover study that is designed to provide continued access to IMCgp100 for eligible participants with advanced melanoma who have previously participated in an IMCgp100 study (parent study).

DETAILED DESCRIPTION:
IMCgp100-401 is a rollover study that is designed to provide continued access to IMCgp100 for eligible participants with advanced melanoma who have previously participated in an IMCgp100 study (parent study). Parent studies that are eligible for participants to continue to receive IMCgp100 in this rollover study must have completed and satisfied its primary endpoints or have been terminated by the Sponsor for reasons other than safety.

Eligible participants will have tolerated IMCgp100 for a minimum of 4 weeks of dosing without significant toxicities that would preclude further dosing in the opinion of the principal investigator or Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is currently participating in an Immunocore-sponsored study of IMCgp100 and is actively receiving IMCgp100. Participant must have fulfilled all required assessments in the parent study (unless the study is being terminated)
2. Participant is currently receiving clinical benefit from the treatment with IMCgp100, as determined by the principal investigator from the parent study
3. Participant has demonstrated compliance with the parent study requirements, as assessed by the principal investigator and participant is able to comply with the necessary visits and assessments as part of the rollover study
4. Written informed consent must be obtained prior to enrolling in the rollover study and receiving the study treatment. If consent cannot be expressed in writing, then the consent must be formally documented and witnessed, ideally via an independent trusted witness

Exclusion Criteria:

1. Participant has been permanently discontinued from any IMCgp100 study or from IMCgp100 treatment in the parent study due to unequivocal progressive disease, unacceptable toxicity, non-compliance to study procedures, withdrawal of consent, or any other reason
2. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin laboratory test
3. Women of child-bearing potential who are sexually active with a non-sterilized male partner, defined as all women physiologically capable of becoming pregnant, unless they are using 2 methods of highly effective contraception from Screening, and must agree to continue using such precautions for 6 months after the final dose of investigational product; cessation of birth control after this point should be discussed with a responsible physician. Highly effective methods include barrier methods, intrauterine devices or hormonal methods. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Women of child-bearing potential must have a negative serum pregnancy test at Screening. Otherwise, female participants must be post-menopausal (no menstrual period for at least 12 months prior to Screening), or surgically sterile
4. Male participants who are not surgically sterile unless they are using a double barrier contraception method from enrollment through treatment and for 6 months following administration of the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Memorial Slone Kettering Cancer Center, New York, New York, United States
- United Kingdom (2):
  - Dept of Oncology & Haematology, Churchill Hospital, Oxford, Oxfordshire
  - Dept of Medical Oncology, Beatson West of Scotland Cancer Centre, Glasgow

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants have tolerated IMCgp100 (77 kDa bi-specific protein) for a minimum of 4 weeks of dosing without significant toxicities that would preclude further dosing in the opinion of the principal investigator or Sponsor.
Pre-assignment Details: Participants were eligible for enrollment in this study from parent studies that have completed and satisfied its primary endpoints or have been terminated by the Sponsor for reasons other than safety.
Groups:
- Regimen 1: IMCgp100 weekly dosing regimen (QW)
Period: Overall Study
Arm/Group | Regimen 1
Started | 3
Completed | 1
Not Completed | 2
Not completed — Ongoing in Survival Follow-up | 2

BASELINE CHARACTERISTICS:
Population: All Patients Enrolled (ENR) set: all participants who provided informed consent for this study.
Groups:
- Regimen 1: IMCgp100 weekly dosing regimen (QW)
  IMCgp100: Bispecific soluble HLA-A2 restricted gp100-specific TCR fused to anti-CD3
Arm/Group | Regimen 1
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events: Number of Participants With Treatment-Emergent Adverse Events
Description: Incidence of adverse events was presented as the number of participants with treatment-emergent adverse events (TEAEs). TEAEs were defined as adverse events (AEs) that started or worsened in severity from the date of first dose of the rollover study (regardless of time) up until 90 days after the last dose of study drug of this rollover study. Participants with multiple events in the same category were counted only once in that category. Participants with events in more than 1 category were counted once in each of those categories. TEAEs indicated considered related to IMCgp100 were determined by the investigator to be possibly related or related to study drug.
Time Frame: Up to 2 years and 4 months
Population: Safety Analysis Set (SAF) includes all participants who have received at least 1 full or partial dose of IMCgp100.
Measure: Number; unit: participants
Arm/Group | Regimen 1
Number analyzed (Participants) | 3
participants
  Any TEAE | 2
  Any TEAE of CTCAE Grade ≥3 | 2
  Any TEAE related to IMCgp100 by Investigator | 2
  Any TEAE of CTCAE Grade ≥3 and related to IMCgp100 | 1
  Any serious TEAE | 0
  Any serious TEAE related to IMCgp100 | 0
  Any TEAE leading to death | 0
  Any TEAE leading to discontinuation of study drug | 0

2. Secondary Outcome: Tolerability: Dose Interruptions by Participant - Number of Cycles
Description: Tolerability of study treatment was assessed by summarizing the number of treatment dose interruptions, characterized in part by number of cycles started and completed in the rollover study (22 days per cycle).
Time Frame: Up to 2 years and 4 months
Population: SAF
Measure: Number; unit: Number of cycles
Groups:
- Participant 4001001 Regimen 1: IMCgp100 weekly dosing regimen (QW)
- Participant 4002001 Regimen 1; Participant 4003001 Regimen 1: MCgp100 weekly dosing regimen (QW)
Arm/Group | Participant 4001001 Regimen 1 | Participant 4002001 Regimen 1 | Participant 4003001 Regimen 1
Number analyzed (Participants) | 1 | 1 | 1
Number of cycles
  Number of cycles started (rollover) | 2 | 26 | 18
  Number of cycles completed (rollover) | 1 | 25 | 17

3. Secondary Outcome: Tolerability: Dose Interruptions by Participant - Duration
Description: Tolerability of study treatment was assessed by summarizing the number of treatment dose interruptions, characterized in part by duration of interruption and treatment.
Time Frame: Up to 2 years and 4 months
Population: SAF
Measure: Number; unit: Days
Groups:
- Participant 4002001 Regimen 1; Participant 4003001 Regimen 1: IMCgp100 weekly dosing regimen (QW)
Arm/Group | Participant 4001001 Regimen 1 | Participant 4002001 Regimen 1 | Participant 4003001 Regimen 1
Number analyzed (Participants) | 1 | 1 | 1
Days
  Duration of IMCgp100 treatment on rollover study | 43 | 728 | 505
  Duration of interruption on rollover study | 0 | 0 | 0
  Duration of IMCgp100 treatment from parent study | 423 | 1156 | 960

4. Secondary Outcome: Tolerability: Dose Reductions by Participant - Actual Total Dose Received
Description: Tolerability of study treatment was assessed by summarizing actual total dose received in micrograms in the rollover study.
Time Frame: Up to 2 years and 4 months
Population: SAF
Measure: Number; unit: Micrograms
Arm/Group | Participant 4001001 Regimen 1 | Participant 4002001 Regimen 1 | Participant 4003001 Regimen 1
Number analyzed (Participants) | 1 | 1 | 1
Micrograms | 350 | 5100 | 3500

5. Secondary Outcome: Tolerability: Dose Reductions by Participant - Dose Intensity
Description: Tolerability of study treatment was assessed by summarizing dose intensity, described as actual dose received/actual duration (micrograms per week) in the rollover study.
Time Frame: Up to 2 years and 4 months
Population: SAF
Measure: Number; unit: Micrograms per week
Arm/Group | Participant 4001001 Regimen 1 | Participant 4002001 Regimen 1 | Participant 4003001 Regimen 1
Number analyzed (Participants) | 1 | 1 | 1
Micrograms per week | 57.0 | 49.0 | 48.5

6. Secondary Outcome: Tolerability: Dose Reductions by Participant - Relative Dose Intensity
Description: Tolerability of study treatment was assessed by summarizing the relative dose intensity, described as the ratio of dose intensity to planned dose/planned duration in the rollover study.
Time Frame: Up to 2 years and 4 months
Population: SAF
Measure: Number; unit: Percent
Arm/Group | Participant 4001001 Regimen 1 | Participant 4002001 Regimen 1 | Participant 4003001 Regimen 1
Number analyzed (Participants) | 1 | 1 | 1
Percent | 100.0 | 100.0 | 100.0

7. Secondary Outcome: Overall Survival Status of All Participants Treated With IMCgp100: Number of Months
Description: This endpoint was used to estimate the overall survival (OS) in participants treated with IMCgp100. OS is defined as the time from the date of first dose of study drug in the parent study until death due to any cause. Any participant not known to have died at the time of analysis was right-censored based on the last recorded date on which the participant was known to be alive, i.e. the latest of (i) the "Date of death or Last contact" (for those participants still alive) on the End of Study electronic case report form page and (ii) "Date patient last known to be alive" on the Survival Follow Up eCRF page. Number of days was then converted to months.
Time Frame: Up to 2 years and 4 months
Population: Full Analysis Set (FAS) comprises all participants assigned to treatment, who received at least 1 full or partial dose of IMCgp100.
Measure: Number; unit: months
Arm/Group | Regimen 1
Number analyzed (Participants) | 3
months
  Baseline to Death: number analyzed (Participants) | 1
  Baseline to Death | 27.0
  Baseline to Study Terminated by Sponsor: number analyzed (Participants) | 1
  Baseline to Study Terminated by Sponsor | 41.0
  Baseline to Alive: number analyzed (Participants) | 1
  Baseline to Alive | 41.0

8. Secondary Outcome: Assessments of Anti-IMCgp100 Antibody Formation: Number of Participants With Anti-IMCgp100 Antibody Formation
Description: The concentration/AE - immunogenicity relationship was explored graphically, and tabulated to characterize a relationship between the changes from screening immunogenicity presence and serum concentration of IMCgp100.
Time Frame: Up to 2 years and 4 months
Population: SAF
Measure: Number; unit: participants
Arm/Group | Regimen 1
Number analyzed (Participants) | 3
participants | 2

ADVERSE EVENTS:
Time Frame: Up to 2 years and 4 months
Description: All participants who received any treatment with IMCgp100 were considered evaluable for safety. All AEs, regardless of study drug relationship, were collected through the 30-day Safety Follow up Period.
Arm/Group | Regimen 1
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen 1 (N=3)
Blepharitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Chills (General disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
ALT increased (Investigations) | 1 (1)
AST increased (Investigations) | 1 (2)
Lipase increased (Investigations) | 1 (5)
White blood cell count decreased (Investigations) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication/presentation (manuscript, abstract or poster) to a journal/scientific meeting is sent to sponsor for review at least 1 month before submission who may delay submission by up to 90 days if it reasonably believes that publication of results may compromise its intellectual property rights or else insist that such data are removed. No single center/groups of centers may publish individually. Publication will not include confidential information without the permission of the sponsor.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT02889861/SAP_000.pdf
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT02889861/Prot_001.pdf